CLINICAL TRIAL: NCT00222677
Title: Aspirin After Six Months or One Year of Oral Anticoagulants for the Prevention of Recurrent Venous Thromboembolism in Patients With Idiopathic Venous Thromboembolism. The WARFASA Study.
Brief Title: Aspirin for the Prevention of Recurrent Venous Thromboembolism
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Of Perugia (Other)
Responsible Party: Principal Investigator, Cecilia Becattini, DR, University Of Perugia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRU-UniPg-01-03
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2011-08-23 (Estimated); Status verified 2011-08

CONDITIONS: Venous Thromboembolism; Deep Venous Thrombosis; Pulmonary Embolism; Atherosclerosis
Keywords: venous thromboembolism; deep vein thrombosis; pulmonary embolism; antithrombotic agents
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism; Atherosclerosis | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: aspirin — 100 mg daily

SUMMARY:
To determine whether aspirin is more effective than placebo for the prevention of recurrent symptomatic venous thromboembolism when given for at least two years after the initial 6-12 month of oral anticoagulant therapy in patients with idiopathic venous thromboembolism

DETAILED DESCRIPTION:
Background

Venous thromboembolism, which includes deep vein thrombosis and pulmonary embolism, is a common disease with an annual incidence of 0.5-1.6 per 1000 in the general population.1-4 Standard treatment with intravenous or subcutaneous heparin or low molecular heparin relayed with oral anticoagulants is highly effective in preventing recurrent episodes of venous thromboembolism.5 However, oral anticoagulant therapy has a number of limitations including an increased risk of major bleeding and the need for laboratory monitoring to adjust dose. Because of these limitations, venous thromboembolism is usually treated with oral anticoagulants for a limited period of time. Anticoagulants are generally discontinued when the risks and inconvenience of remaining on treatment outweigh the risk of recurrent venous thromboembolism. Indeed, recent studies showed that after discontinuation of anticoagulant treatment, the risk of recurrent venous thromboembolism remains high in patients with idiopathic venous thromboembolism.

Recently, four major randomized trials have evaluated extended-duration treatment with oral anticoagulants in patients with venous thromboembolism. In each of these trials more than 90% of recurrences occurred after oral anticoagulants had been discontinued 6-9. The rate of recurrence after discontinuation of oral anticoagulants was similar in patients assigned long-term therapy compared with short-term therapy (about 15% in the 2-3 years after warfarin discontinuation) which indicates that although oral anticoagulants are highly effective to prevent recurrence, it have no impact on the natural history of idiopathic venous thromboembolism. Taken together, these data suggest that effective therapy should be continued indefinitely in patients with idiopathic venous thromboembolism if recurrence is to be avoided. Indeed, once oral anticoagulants are discontinued, there are currently no established safe and effective alternatives to prevent recurrence in patients with idiopathic venous thromboembolism. However, the long-term use of oral anticoagulants is not only inconvenient because of the need for close laboratory monitoring but also is constrained by an increased risk of major bleeding, including fatal and intracranial bleeding. In randomized trials of extended-duration oral anticoagulants (target INR 2.0-3.0) for the treatment of venous thromboembolism,6-9 the annual incidence of intracranial bleeding was 0.3%, major bleeding 3%, and the case-fatality rate of major bleeding approximately 10%. In addition, 5-15% of patients experienced minor bleeding each year. These data highlight the need to identify simple, safe, effective, and widely applicable strategies for the long-term prevention of recurrent deep vein thrombosis or pulmonary embolism in patients with idiopathic venous thromboembolism.

About 3% of patients with venous thromboembolism experience an arterial cardiovascular event (myocardial infarction, stroke, sudden otherwise unexplained death) in the 2-3 years after the first episode of venous thromboembolism10. The long-term use of oral anticoagulants could potentially prevent these adverse events. Barriers to the more widespread appropriate use of oral anticoagulants include physician concerns regarding the risk of bleeding, particularly in the elderly, as well as the need for close monitoring and regular blood tests to measure the INR. A simple, safe, effective, and widely applicable pharmacological approach is needed for the prevention of these events.

The clinical utility of aspirin in the management of venous thromboembolism is a matter of debate. The Pulmonary Embolism Prevention Study 11 demonstrated that 35 days of low-dose aspirin (160 mg daily) compared with placebo reduced the risk of symptomatic venous thromboembolism, including fatal pulmonary embolism, by about one-third (RRR 36%, 95% CI: 19-50%, p=0.0003) in patients undergoing emergency surgery for hip fracture or elective joint arthroplasty. There was no excess of fatal or intracranial bleeding. In the Heart and Estrogen/progestin Replacement Study (HERS)12 2800 postmenopausal women with coronary artery disease were randomized to hormonal replacement therapy or placebo. A secondary analysis showed that the use of aspirin was independently associated with a 50% reduction (95% CI: 20-80%) in risk of venous thromboembolism during an average of 4.1 years of follow-up. Taken together, these data suggest that aspirin reduces the risk of a first episode of venous thromboembolism by about one-quarter (i.e., 25% risk reduction).

A systematic overview including more than 8000 patients from randomized trials on antiplatelet primary thromboprophylaxis suggested that antiplatelet therapy was effective to prevent deep vein thrombosis and pulmonary embolism in high risk patients (Antiplatelet Trialists' Collaboration).13 Antiplatelet therapy was associated with a relative risk reduction [RRR] of 39%; (p=0.00001) in the incidence of venous thromboembolism in high-risk medical patients or undergoing orthopedic or general surgery. There was no excess in cerebral or fatal bleeding.

The European Stroke Prevention Study 2 (ESPS 2)14 evaluated the efficacy and safety of aspirin, dipyridamole (extended-release preparation), or aspirin and dipyridamole, versus placebo, for the secondary prevention of ischemic stroke in 6,600 patients. Prespecified secondary analyses found that aspirin resulted in a 30% reduction in venous thromboembolism.

Bleeding, particularly within the gastrointestinal tract, is the only important side effect of low-dose aspirin therapy in patients that are not already known to be aspirin intolerant (e.g., allergy). Long term, low-dose aspirin therapy (i.e., 160 mg per day), is associated with about a two-fold increase in the risk of bleeding.15-17 This increase of bleeding is small in patients without known contraindications to aspirin. Evidences from randomized trials of aspirin in asymptomatic subjects, patients with vascular risk factors, or patients with a past history of vascular disease (more than 250,000 patient-years of follow-up), showed an absolute excess of major bleeding with aspirin from 0.3 to 1.7 episodes per 1000 patient-years, equivalent to an absolute risk of 1 event for every 1000 patients treated.15 Increasing doses of aspirin, even within the range of 100-300 mg per day, were associated with an increasing risk of gastrointestinal bleeding, with the lowest risk occurring in patients receiving 100 mg daily.15;18-19

In summary, aspirin could achieve a risk reduction of 30 to 40 episodes of deep vein thrombosis or pulmonary embolism for every 1000 patients treated, at a cost of 1 bleed requiring transfusion in high-risk patients with idiopathic venous thromboembolism. Aspirin is simple to administer and does not require laboratory monitoring.

In the present study we propose to evaluate the use of low-dose aspirin for the prevention of recurrent venous thromboembolism in patients with previous idiopathic venous thromboembolism who have received initial 6-month treatment with oral anticoagulants.

ELIGIBILITY:
Inclusion Criteria:

* first episode of symptomatic, objectively confirmed idiopathic proximal deep vein thrombosis and/or pulmonary embolism;
* initial treatment with unfractionated heparin or low-molecular-weight heparin (or effective alternative) followed by a vitamin K antagonist (target INR 2.0-3.0). All patients will receive 6 or 12 months of oral anticoagulant treatment. Patients initially treated with thrombolytic therapy who received warfarin therapy are eligible for inclusion.

Exclusion Criteria:

* permanent risk factors for venous thromboembolism: patients known to have antiphospholipid antibodies or lupus anticoagulant (based on local laboratory criteria) or to have homozygous factor V Leiden or homozygous prothrombin G21210A or heterozygous factor V Leiden plus heterozygous prothrombin G21210A or antithrombin III deficiency; patients with active malignancy
* temporary risk factors for venous thromboembolism
* any recurrence of venous thromboembolism or bleeding episode during the established 6-month period of oral anticoagulant treatment
* allergy or intolerance of aspirin
* clear indication for aspirin or other anti-platelet therapy (e.g. clopidogrel, ticlopidine)
* clear indication for long-term anticoagulant therapy (e.g. recurrent idiopathic venous thromboembolism, prosthetic heart valve)
* treatment with non-selective COX-1/2 non-steroidal anti-inflammatory drugs
* life expectancy less than 6 months
* active bleeding or at high risk of bleeding (gastrointestinal bleeding within the past 12 months; endoscopic diagnosis of peptic ulcer disease or ulcerative esophagitis within the past 6 months unless there is documented endoscopic evidence of healing; intracranial bleeding within the past year; known bleeding diathesis)
* anticipated non-adherence to study medications
* inability to attend follow up because of geographic inaccessibility
* failure to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2004-05; Primary Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
recurrence of VTE and/or VTE related death | at least 24 months per patient

SECONDARY OUTCOMES:
recurrent VTE+ death; cardiovascular events, bleeding events, critical ischemia of the lower limbs, mesenteric infarction, all cause mortality and newly diagnosed cancer | at least 24 months per patient

CONTACTS AND LOCATIONS:
Overall Officials: Giancarlo Agnelli, MD, Study Chair — Department of Internal Medicine - University of Perugia; Cecilia Becattini, MD, Study Director — Department of Internal Medicine - University of Perugia; Paolo Prandoni, PhD, Study Director — University of Padova
Locations (15):
- Department of Internal Medicine - University of Vienna, Vienna, Austria
- Italy (14):
  - Unità di Aterosclerosi e Trombosi -Casa Sollievo della Sofferenza, San Giovanni Rotondo, FG
  - Divisione di Ematologia, Dipartimento di Medicina Interna - Università di Milano-Bicocca, Monza, Milano
  - Angiologia - Osp. Garibaldi - Piazza S. Maria del Gesù, 7, Catania
  - UO di Medicina 'Valentini' - PO 'Annunziata', Cosenza
  - Angiologia - Ospedale di Faenza, Faenza
  - Divisione Medica II - Ospedale Galliera, Genova
  - Centro Emofilia e Trombosi - Ospedale Maggiore di Milano IRCCS, Milan
  - Clinica Medica II - Università di Padova, Padua
  - Unità malattie tromboemboliche ed emorragiche - Azienda universitaria Policlinico, Palermo
  - Internal and Cardiovascular Medicine - University of Perugia, Perugia
  - Medicina Interna I - Arcispedale S. Maria Nuova, Reggio Emilia
  - Divisione Medica I, Ospedale Cà Foncello, Treviso
  - Medicina d'Urgenza - Ospedale Cattinara, Trieste
  - Department of Medicina Interna e Terapia Medica, Università dell'Insubria, Varese

REFERENCES:
- [Derived] Flumignan CD, Nakano LC, Baptista-Silva JC, Flumignan RL. Antiplatelet agents for the treatment of deep venous thrombosis. Cochrane Database Syst Rev. 2022 Jul 25;7(7):CD012369. doi: 10.1002/14651858.CD012369.pub2. PMID 35876829
- [Derived] Becattini C, Agnelli G, Schenone A, Eichinger S, Bucherini E, Silingardi M, Bianchi M, Moia M, Ageno W, Vandelli MR, Grandone E, Prandoni P; WARFASA Investigators. Aspirin for preventing the recurrence of venous thromboembolism. N Engl J Med. 2012 May 24;366(21):1959-67. doi: 10.1056/NEJMoa1114238. PMID 22621626